CLINICAL TRIAL: NCT04160364
Title: Gender Dysphoria in Children and Adolescents : Parents' Perspectives
Acronym: GeDyPar
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PI204
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-07

CONDITIONS: Gender Dysphoria
Keywords: children; adolescents; parents
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: qualitative study — qualitative research via guided interview

SUMMARY:
Gender dysphoria is defined as a persistent incongruence between an experienced gender and the assigned sex at birth Transgender and gender nonconforming persons desire to modify their appearance to be consistent with their self-identified gender identities. In non-binary people, contrary to binary transgender persons, self-identified gender identities do not fit the classical pattern male/female.

During the last decennium, an increase in the number of young subjects, especially children and adolescents, referred to gender identity centres has been observed. A new nosological entity "rapid-onset gender dysphoria in adolescents and young adults" has recently been described in the literature, whose etiology has not been well understood.

This growing demand of adolescents and young adults observed in the recent years is not well understood.

ELIGIBILITY:
Inclusion Criteria:

* be a parent of a child <18 years followed in the endocrinology department of the University Hospital of Nancy for gender dysphoria
* be in stable couple
* both parents agree to participate
* capacity to communicate in French
* Person who has received complete information on the organization of the research and who agreed to the exploitation of the data

Exclusion Criteria:

* Refusal to participate
* Inability to be physically, psychologically or linguistically involved in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be proposed to parents of transgender children <18 years of age followed in the endocrinology, diabetology and nutrition department of the University Hospital of Nancy on the occasion of the regular follow-up visit at the outpatient clinic ( consecutive recruitment).
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
thematic analysis | one year
  The recorde material will be coded using descriptive codes. Conceptual notes will be written, through processes of condensation, comparison and abstracting the initial notes.
  Connections between notes will be noted and synthesized, and emergent themes will be developed.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Feigerlova, MD,PhD, Principal Investigator — University Hospital of Nancy, France
Locations (1):
- University Hospital of Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No
Not planned